CLINICAL TRIAL: NCT00942539
Title: Midazolam Sedation for Neonatal Lumbar Puncture in the Emergency Department: A Randomized Controlled Trial
Brief Title: Midazolam Sedation for Neonatal Lumbar Puncture
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, i_shavit, Pediatric Emergency Department director, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2958CTIL
Record Dates: First submitted 2009-07-18; First posted 2009-07-21 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2010-07

CONDITIONS: Pain; Anxiety
Keywords: Neonates
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Midazolam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Midazolam (Experimental): Administration of Midazolam prior Lumbar Puncture
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — Intravenous infusion of 0.05 mg/kg of Midalolam

SUMMARY:
Lumbar puncture is one of the most common painful procedures performed on neonates in the Emergency Department (ED). The investigators will study in a randomized controlled trial, the efficacy of intravenous administration of a single dose of Midazolam in reducing pain and anxiety in neonates undergoing lumbar puncture in the ED, as well as the rate of adverse sedation reactions. The investigators hypothesize that compared with placebo, single dose Midazolam would significantly decrease pain and anxiety and will have low rate of adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) score I, II
* Post natal age ≤ 30 days
* Fasting of at least 2 hours before the procedure

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) score III or greater
* Gestational age of 37 weeks or younger
* Congenital disease or defect
* Any medication provided by the caregiver prior ED admission
* Fasting of less than 2 hours

Ages: 3 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The Simplified Neonatal Facial Coding System will be used for assessment of pain. Scoring will be composed from four specific facial actions (brow bulge, nasolabial furrow, eye squeeze, and open mouth) and the presence or absence of crying | 20 seconds prior lumbar puncture, during needle insertion, and 20 seconds post insertion

SECONDARY OUTCOMES:
Physician's level of satisfaction from the procedural conditions | Five minutes post successful LP
LP Success rate | Five minutes post successful LP
Adverse sedation reactions | During procedure and during recovery phase

CONTACTS AND LOCATIONS:
Overall Officials: Itai Shavit, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel